CLINICAL TRIAL: NCT05594953
Title: Outcomes Using MARS: A Single Center Experience
Brief Title: Outcomes Using MARS for Patients With ALF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 075.HEP.2020.D
Record Dates: First submitted 2022-02-03; First posted 2022-10-26 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-07

CONDITIONS: Alcoholic Hepatitis; Acute Liver Failure
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Failure, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective chart review will be conducted on patients at Methodist Dallas Medical Center, meeting the inclusion criteria from January 1, 2019 to December 15, 2020 to determine the transplant free survival and overall survival and other secondary outcome measures.

DETAILED DESCRIPTION:
Retrospective chart review will be conducted on patients at Methodist Dallas Medical Center, meeting the inclusion criteria from January 1, 2019 to December 15, 2020 to determine the transplant free survival and overall survival and other secondary outcome measures. Patient's charts will be accessed on EPIC by the PI or delegated study personnel. The investigator's anticipate completion of this study by January 31, 2022.

ELIGIBILITY:
Inclusion Criteria:

• The patient was diagnosed with: Alcoholic hepatitis; AoCLF; OR Acute fulminant liver failure

• The patient underwent at least one round of dialysis using plasma exchange or MARSTM

Exclusion Criteria:

* Patient not meeting the inclusion criteria will be excluded.

All patients who underwent MARS at MDMC will be included in the study population.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients meeting the inclusion criteria (Alcoholic hepatitis, AoCLF; or ALF who underwent at least one round of dialysis using plasma exchange or MARS from January 1, 2019 to December 15, 2020 will be included in the analysis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival mortality | Rate at 30 days
  transplant will be measured by date of death, and discharge
Difference in Demographics | Rate at 30 days
  co-morbidities, etiology of liver failure between those treated with MARS vs. controls
Improvement in Transplant | Rate at 30 days
  Determine whether treatment with MARS can help facilitate improvement in HE, LOS, and ICU duration.

SECONDARY OUTCOMES:
Demographics | January 1, 2019 to January 31, 2022
  age (years), gender (male/female), race (Caucasian, black, Hispanic, Asian, other), BMI (kg/m2)
Hepatorenal syndrome | (in hospital [date of death or discharge or transplant]) and at 30 days
  Y/N
Need for vasopressor support | (in hospital [date of death or discharge or transplant]) and at 30 days
  Y/N
Sepsis (as measured by by QSOFA criteria): | (in hospital [date of death or discharge or transplant]) and at 30 days
  Y/N
Need for CRRT as documented in the chart: | (in hospital [date of death or discharge or transplant]) and at 30 days
  Y/N
ICU duration | date of ICU admission and date of discharge (or death)
  days of date of ICU duration
long term dialysis | (in hospital [date of death or discharge or transplant]) and at 30 days
  Need for long term dialysis (Y/N)

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Mantry, MD, Principal Investigator — Methodist
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States